CLINICAL TRIAL: NCT05617950
Title: Salicylic Acid Versus Cryotherapy for the Treatment of HPV1-induced Plantar Warts: a Randomized Controlled Trial
Brief Title: Salicylic Acid Versus Cryotherapy for the Treatment of HPV1-induced Plantar Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The 306 Hospital of People's Liberation Army (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 306PLA-005
Record Dates: First submitted 2022-11-01; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Salicylic Acid; Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- salicylic acid (Experimental): 30% salicylic acid
  Interventions: Other: salicylic acid
- cryotherapy (Active Comparator): liquid nitrogen
  Interventions: Other: cryotherapy

INTERVENTIONS:
Other: salicylic acid — Salicylic acid is applied once daily by the patients (or parents) for a maximum of 12 weeks.
  Arms: salicylic acid
Other: cryotherapy — Cryotherapy is delivered by a technician up to a maximum of four treatments 3 weeks apart.
  Arms: cryotherapy

SUMMARY:
To evaluate whether salicylic acid was superior to cryotherapy for plantar warts

DETAILED DESCRIPTION:
Patients with plantar warts were randomized equally to receive salicylic acid or cryotherapy. Cryotherapy is delivered by a technician up to a maximum of four treatments 3 weeks apart. Thirty percent of salicylic acid is applied once daily by the patient (or parent) for a maximum of 12 weeks. The primary outcomes were the cure rates at 12 weeks; secondary outcomes included time to clearance of warts, patient satisfaction with the treatment and treatment-related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HPV1-induced plantar warts.
* Total number of warts is ≤5.
* Aged 12 years or older.

Exclusion Criteria:

* Patients are currently participating in another trial for the treatment of plantar warts.
* Patients had received two or more consecutive sessions of cryotherapy, with an interval of no more than 4 weeks (The history of salicylic acid treatment was not considered as criteria for exclusion because high concentration salicylic acid is not commercially available in Chinese mainland).
* Patients have taken immunosuppressant drugs (such as oral corticosteroids) during the past three months.
* Patients have impaired healing eg due to diabetes, vitamin A deficiency, hyperthyroidism and hypothyroidism.
* Patients have autoimmune diseases (such as systemic lupus erythematosus, dermatomyositis, scleroderma or other diseases).
* Patients are pregnant or ready for pregnancies or breast-feeding.
* Patients have cold intolerance (such as cold urticaria, cryoglobulinaemia, cold agglutinin syndrome or Raynaud's syndrome).
* Patients have local pain intolerance.
* Patients have local hypoesthesia.
* Patients are unable to tolerate salicylic acid or cryotherapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
cure rate at 12 weeks | 12 weeks since the initial treatment
  A patient was considered to be cured if all warts were no longer visible and could not be palpated anymore.

SECONDARY OUTCOMES:
time to clearance of warts | 12 weeks since the initial treatment
  The time from treatment initiation until clearance of all warts
patient satisfaction with the treatment | 12 weeks since the initial treatment
  Patient satisfaction was rated on a 5-point scale (from very happy to very unhappy)
treatment-related adverse events | 12 weeks since the initial treatment
  Some adverse effects, including pain, swelling, blisters, hemorrhagic bullae, bruising, and skin breakdown, were recorded by the patients, whereas others, including secondary bacterial infection, hyperpigmentation, hypopigmentation, and scarring were evaluated by a dermatologist

CONTACTS AND LOCATIONS:
Overall Officials: Shichao Lu, MD, Principal Investigator — The 306 Hospital of People's Liberation Army